CLINICAL TRIAL: NCT02835196
Title: Optical Elastography of Systemic Sclerosis Skin
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Shervin Assassi, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-16-0383; PR150338 (Other Grant/Funding Number: Congressionally Directed Medical Research Program)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Ergonomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin punch biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Optical Elastography Assessment of Skin Thickness
  Interventions: Device: Optical Elastography
- Visual Assessment of Skin Thickness
  Interventions: Other: Visual Assessment

INTERVENTIONS:
Device: Optical Elastography — To image skin thickness, Optical Coherence Elastography (OCE)-scanning of 6 body surface areas will be preformed using the Phase-Stabilized Swept Source Optical Coherence Elastography (PhS-SSOCE) system.
  Groups: Optical Elastography Assessment of Skin Thickness
Other: Visual Assessment — Skin thickness will be visually assessed clinically in 6 body surface areas using the the modified Rodnan Skin Score (mRSS). The mRSS uses a 0-3 scale, where 0 = normal, 1= mild thickness, 2 = moderate thickness, and 3 = severe thickness
  Groups: Visual Assessment of Skin Thickness

SUMMARY:
The goal of this study is to develop a new way to assess skin thickness in patients with scleroderma (systemic sclerosis). The study will test how well a new imaging method called optical coherence elastography (OCE) compares to the current clinical method used to estimate skin thickness, the modified Rodnan Skin Score (mRSS).

ELIGIBILITY:
Inclusion Criteria for scleroderma patients:

* meet the 2013 American College of Rheumatology and the European League Against Rheumatism (ACR/EULAR) criteria for systemic sclerosis with limited or diffuse cutaneous involvement

Exclusion Criteria:

* have another skin disease other than systemic sclerosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Skin optical elastography (OCE) scan score | Baseline

SECONDARY OUTCOMES:
Skin thickness as assessed by Modified Rodnan Skin Score (mRSS) | Baseline
Fibrosis score as assessed by forearm skin punch biopsy | Baseline
  A score based on histological findings of skin punch biopsy will be calculated. There some minor risk involved with skin biopsy procedure.
Disability as assessed by the Scleroderma Health Assessment Questionnaire | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shervin Assassi, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No